CLINICAL TRIAL: NCT04481048
Title: Antioxidant Therapy With N-acetylcysteine for Motor Behavior and/or Learning in Children With Neurofibromatosis Type 1
Brief Title: Antioxidant Therapy With N-acetylcysteine for Children With Neurofibromatosis Type 1
Acronym: DoDNAC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-0412
Record Dates: First submitted 2020-05-15; First posted 2020-07-22 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-08

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Acetylcysteine; Inhalation

STUDY DESIGN:
Intervention Model Description: This is a phase II, double blind, placebo-controlled clinical trial with the goal to explore safety, tolerability, and efficacy of N-acetylcysteine (NAC).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In order to preserve the double-masking of the trial, only the investigation pharmacy will be unmasked. Both treatments (NAC and placebo) will be distributed from the investigational pharmacy. Except for the pharmacist, all staff will be blinded to the treatment sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- N-Acetylcysteine (NAC) (Experimental): Each subject will be dosed with approximately 70 mg/kg/day of NAC for 8 weeks. To facilitate drug compounding, three tiers of drug dose will be administered based on body weight as described in Table 3.
  Table 3: NAC Dosing Participant's weight (kg) Dose (BID) < 20 700 mg 21-39 1050 mg > 40 1350 mg
  *Max dose not to exceed 2700mg/day (1350mg BID)
  Interventions: Drug: N-Acetyl cysteine
- Placebo (Placebo Comparator): Each subject will be dosed with placebo for 8 weeks.
  Interventions: Other: Placebo
- Single Visit/Non-Treatment Arm (No Intervention): Based on preliminary data, an additional "Single visit, non-treatment" cohort will include 40 individuals with NF1 for a single "biomarker" study visit. These individuals will undergo motor function (PANESS) and brain-based measures (TMS, MRI-MRS, DTI) as biomarkers of impaired executive function (ADHD-RS; BRIEF-2; TOVA) but will not be assigned to receive NAC/Placebo.

INTERVENTIONS:
Drug: N-Acetyl cysteine — Eight (8) weeks of treatment with an FDA approved medication, N-acetylcysteine (NAC).
  Other Names: •Chemical Name: Cysteine, N-acetyl-, L; •Commercial Name(s): Acetein; Acetadote, Acetylcysteine; Airbron; Broncholysin; Fluimucetin; Fluimucil; Inspir; Mucofilin; Mucomyst; Mucosolvin; NAC; Paravolex; Respaire; •Synonym:L-alpha-acetamido-beta-mercaptopropionic acid; Mercpaturic acid; N-Acetyl-3-mercaptoalanine; N-Acetylcysteine
  Arms: N-Acetylcysteine (NAC)
Other: Placebo — Eight (8) weeks of treatment with placebo.
  Arms: Placebo

SUMMARY:
Children with neurofibromatosis type 1 (NF1) commonly suffer from the effects of cognitive, behavioral, and motor impairments. At present, there is no specific treatment for this NF1 complication. In this project, the investigators will assess the safety and clinical benefit of N-acetylcysteine (NAC) as a pharmacological intervention in children with NF1. This drug choice is based on the recent findings from mouse models to study the central nervous system manifestations of NF1 at Cincinnati Children's Hospital Medical Center (CCHMC). These findings revealed a role for myelin-forming oligodendrocytes in the control of nitric oxide synthases (NOS) and their product, nitric oxide (NO), in maintenance of brain structure and function, including regulation of behavior and motor control. Treating these mice with NAC corrected cellular and behavioral abnormalities. This data from animal models of NF1 along with uncontrolled clinical observations in children with NF1 suggest that the antioxidant compound, NAC, may reduce these impairments. Therefore, the investigators propose performing a single center double-blind placebo controlled, prospective, Phase II study to explore safety, tolerability, and efficacy of NAC on motor behavior and/or learning in children with NF1 aged 8 through 16 years old. Participants will be carefully monitored for side effects. Primary and secondary outcome measures will be administered at baseline, follow-up, and post-treatment.

DETAILED DESCRIPTION:
This is a phase II clinical trial with the goal to explore safety, tolerability, and efficacy of NAC on motor behavior in children with NF1 aged 8 through 16 years old. The investigators hypothesize that NAC therapy will improve motor function evaluated by the PANESS scale. This is based on studies demonstrating that NAC significantly improved impairments in the animal model of NF1. The investigators will also analyze NAC effects on attention deficit and impulsivity in children with NF1.

This study will also help develop novel predictive biomarkers of response to neurocognitive therapies in patients with NF1 which are needed to evaluate treatment outcomes.

The investigators will gain information in children with NF1 about possible clinical benefit of anti-oxidant treatment and to develop and evaluate quantitative brain-based and blood biomarkers relating to presence of NF1, symptom severity, and response to antioxidant therapy. Clinically, 50 percent of children with NF1 are underperforming or failing at school. This frequently leads to decreased educational attainment and fewer opportunities as adults. An important first step was preliminary work using the PANESS scale and Transcranial Magnetic Stimulation (TMS)-evoked Short Interval Cortical Inhibition (rSICI) in children with NF1. The investigators propose to develop and extend understanding of NF1-related motor and learning behavior in response to antioxidant therapy with NAC. The purpose of the present study is to 1) evaluate tolerability, safety, and clinical benefit of NAC in this double-blind placebo controlled study using the motor function scale (PANESS); 2) to evaluate the effects of NAC on measures of NF1 neurocognitive symptomatology (ADHD/impulsive symptoms, executive function, working memory); and 3) to determine if TMS measurement (SICI) in children with NF1 will correlate with clinical effects of NAC treatment and evaluate utility of advanced brain imaging and spectroscopy measurements in children with NF1, and effects of NAC therapy.

The investigators propose to study 58 children with NF1, ages 8-16 years, at baseline and after completion of 8 weeks of treatment with NAC, followed by a washout period of 4 weeks.

The investigators believe this work has the potential to lay groundwork for future use of relevant biomarkers for treatment and outcomes research for NF1 as well as other biologically similar conditions, collectively designated the "RASopathies" (due to involvement of the RAS family of proteins) and ultimately to guide development of more effective treatments based on disease pathophysiology.

STUDY OBJECTIVE:

NAC Trial at Cincinnati Children's Hospital Medical Center (CCHMC) The investigators propose performing a single center randomized double-blind placebo controlled, prospective, Phase II study to explore safety, tolerability, and efficacy of NAC on motor behavior in children with NF1 aged 8 through 16 years old.

Hypothesis:

The investigators hypothesize that NAC therapy will improve motor function evaluated by the PANESS scale. This is based on studies demonstrating that NAC significantly improved impairments in the animal model of NF1. The investigators will also analyze NAC effects on attention deficit and impulsivity in children with NF1.

Specific Aim:

The primary outcome of this study is to characterize the effects of NAC treatment on motor function in children and adolescents with NF1 using the PANESS. The investigators hypothesize that motor function scores rated with the PANESS scale will improve after treatment with NAC.

Secondary Aims:

1. To evaluate the effects of NAC on measures of NF1 neurocognitive symptomatology (ADHD/impulsive symptoms, executive function, working memory), the investigators will use Response Evaluation in Neurofibromatosis and Schwannomatosis (REiNS) committee recommended assessments tools DuPaul ADHD rating scale (ADHD-RS), Behavioral Rating Inventory of Executive Function second edition (BRIEF-2), Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) subtests, and Test of Variables of Attention (TOVA).
2. To determine if TMS measurement (SICI) in children with NF1 will correlate with clinical effects of NAC treatment.
3. To quantify microstructural properties of brain tissue based on water diffusion, glutathione GSH concentrations, and gamma-aminobutyric acid (GABA) concentration using brain magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) in children with NF1. This will allow for regional correlation between imaging, spectroscopy and neuropsychometric outcomes. The investigators will also determine if these magnetic resonance based outcomes correlate with clinical effects of NAC treatment.
4. To evaluate safety and tolerability of NAC in children with NF1.

ELIGIBILITY:
Inclusion Criteria ѱ:

You can be in this study if you have any of the following:

1. Males and females older than 8 years and younger than 16 years old
2. Has a diagnosis of NF1 (neurofibromatosis type 1)
3. Has an abnormal PANESS score
4. Has an IQ (intelligence quotient) at or above 70
5. Participants on stimulant or any other psychotropic medication should stay on a stable dose (no change in dose) for at least 30 days before entering the study and maintain that dose while in the study

Exclusion Criteria:

You cannot be in this study if you have any of the following:

1. Younger than 8 years or older than 16 years ѱ
2. Do not have a diagnosis of NF1 ѱ
3. IQ below 70 ѱ
4. Had a dose change of any stimulant or psychotropic medication in the last month (30 days) ѱ
5. Are being treated with chemotherapy or had chemotherapy in the last 6 months
6. Have epilepsy ѱ
7. High risk of upper gastrointestinal (GI, the stomach and the small and large intestine) hemorrhage (bleeding). Examples: presence of esophageal varices or peptic ulcers
8. Active intracranial lesions (abnormality found on brain imaging such as an MRI) (stable low-grade glioma is acceptable) or epilepsy diagnosis ѱ
9. Have Major Depression, Bipolar Disorder, Conduct Disorder, Adjustment Disorder, other major Anxiety Disorders, or other developmental psychiatric diagnoses, based on history. ADHD is OK
10. For females, pregnancy
11. Is currently using antidepressants, dopamine blocking agents, or mood stabilizers
12. Have any of the following medical devices: implanted brain stimulator, vagal nerve stimulator, VP (ventriculoperitoneal) shunt, cardiac pacemaker, or implanted medication port ѱ
13. Asthma (bronchospasm has been reported as occurring infrequently and unpredictably when NAC is used as a mucolytic agent)
14. Current use of MEKINIST (MEK-inhibitor) or use within 30 days

ѱ Indicates Inclusion/Exclusion Criteria for the treatment- and non-treatment cohorts (no mark indicates exclusion requirements for the 12-week treatment-cohort only).

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Motor Function Measured by Physical and Neurological Examination for Subtle Signs (PANESS) | through 12 weeks (at weeks 0, 8, and 12)
  Characterize effects of NAC treatment on motor function in kids with NF1 using the Physical and Neurological Examination for Subtle Signs (PANESS). This is a validated scale that consistently demonstrates significant impairments in children with ADHD, and which preliminary data suggest may demonstrate more extreme problems in children with NF1 than age-matched healthy controls (unpublished data from CCHMC). The investigators hypothesize that motor function scores rated with the PANESS scale will improve after treatment with NAC. The range of this scale is 0-119, higher scores correlate with symptom severity (worse outcome).

SECONDARY OUTCOMES:
Change from Baseline in ADHD Symptoms as Reported via Parent/Teacher Surveys | through 12 weeks (at weeks 0, 8, and 12)
  Characterize effects of NAC treatment on ADHD symptoms in children with NF1. The investigators hypothesize that ADHD attention and hyperactive/impulsive symptoms, rated with the DuPaul Diagnostic and Statistical Manual Diploma in Social Medicine (DSM-5) based clinical rating scales, will improve after treatment with NAC. The range of this scale is 0-56, higher scores correlate with symptom severity (worse outcome).
Change from Baseline in Motor Function and Physiology Measured by Transcranial Magnetic Stimulation (TMS) | through 12 weeks (at weeks 0, 8, and 12)
  Describe the function and physiology of the motor system using Transcranial Magnetic Stimulation (TMS) as a possible disease biomarker of NF1. Preliminary measures in an NF1 population also show abnormalities similar to established findings in ADHD. The investigators hypothesize that children with NF1 will have significantly less motor cortex inhibition using TMS measurements, and these measures will improve ("normalize") upon NAC treatment. The investigators will compare to our internal age-matched healthy controls at Cincinnati Children's.
Change from Baseline in Microstructural Properties of Brain Tissue Visualized by Magnetic Resonance Imaging (MRI) | through 12 weeks (at weeks 0, 8, and 12)
  To quantify microstructural properties of brain tissue based on water diffusion, glutathione GSH concentrations, and gamma-aminobutyric acid (GABA) concentration using brain magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) in children with NF1. This will allow for regional correlation between imaging, spectroscopy and neuropsychometric outcomes. We will also determine if these magnetic resonance based outcomes correlate with clinical effects of NAC treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Gilbert, MD MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acosta MT, Gioia GA, Silva AJ. Neurofibromatosis type 1: new insights into neurocognitive issues. Curr Neurol Neurosci Rep. 2006 Mar;6(2):136-43. doi: 10.1007/s11910-996-0036-5. PMID 16522267
- [Background] Ballester R, Marchuk D, Boguski M, Saulino A, Letcher R, Wigler M, Collins F. The NF1 locus encodes a protein functionally related to mammalian GAP and yeast IRA proteins. Cell. 1990 Nov 16;63(4):851-9. doi: 10.1016/0092-8674(90)90151-4. PMID 2121371
- [Background] Rosser TL, Packer RJ. Neurocognitive dysfunction in children with neurofibromatosis type 1. Curr Neurol Neurosci Rep. 2003 Mar;3(2):129-36. doi: 10.1007/s11910-003-0064-3. PMID 12583841
- [Background] Casnar CL, Janke KM, van der Fluit F, Brei NG, Klein-Tasman BP. Relations between fine motor skill and parental report of attention in young children with neurofibromatosis type 1. J Clin Exp Neuropsychol. 2014;36(9):930-43. doi: 10.1080/13803395.2014.957166. Epub 2014 Oct 6. PMID 25284746
- [Background] Walsh KS, Janusz J, Wolters PL, Martin S, Klein-Tasman BP, Toledo-Tamula MA, Thompson HL, Payne JM, Hardy KK, de Blank P, Semerjian C, Gray LS, Solomon SE, Ullrich N; REiNS International Collaboration. Neurocognitive outcomes in neurofibromatosis clinical trials: Recommendations for the domain of attention. Neurology. 2016 Aug 16;87(7 Suppl 1):S21-30. doi: 10.1212/WNL.0000000000002928. PMID 27527646
- [Background] Acosta MT, Bearden CE, Castellanos FX, Cutting L, Elgersma Y, Gioia G, Gutmann DH, Lee YS, Legius E, Muenke M, North K, Parada LF, Ratner N, Hunter-Schaedle K, Silva AJ. The Learning Disabilities Network (LeaDNet): using neurofibromatosis type 1 (NF1) as a paradigm for translational research. Am J Med Genet A. 2012 Sep;158A(9):2225-32. doi: 10.1002/ajmg.a.35535. Epub 2012 Jul 20. PMID 22821737
- [Background] Pride N, Payne JM, Webster R, Shores EA, Rae C, North KN. Corpus callosum morphology and its relationship to cognitive function in neurofibromatosis type 1. J Child Neurol. 2010 Jul;25(7):834-41. doi: 10.1177/0883073809350723. Epub 2010 Feb 8. PMID 20142468
- [Background] Wang Y, Kim E, Wang X, Novitch BG, Yoshikawa K, Chang LS, Zhu Y. ERK inhibition rescues defects in fate specification of Nf1-deficient neural progenitors and brain abnormalities. Cell. 2012 Aug 17;150(4):816-30. doi: 10.1016/j.cell.2012.06.034. PMID 22901811
- [Background] Karlsgodt KH, Rosser T, Lutkenhoff ES, Cannon TD, Silva A, Bearden CE. Alterations in white matter microstructure in neurofibromatosis-1. PLoS One. 2012;7(10):e47854. doi: 10.1371/journal.pone.0047854. Epub 2012 Oct 19. PMID 23094098
- [Background] Gilbert DL, Isaacs KM, Augusta M, Macneil LK, Mostofsky SH. Motor cortex inhibition: a marker of ADHD behavior and motor development in children. Neurology. 2011 Feb 15;76(7):615-21. doi: 10.1212/WNL.0b013e31820c2ebd. PMID 21321335
- [Background] Chen TH, Wu SW, Welge JA, Dixon SG, Shahana N, Huddleston DA, Sarvis AR, Sallee FR, Gilbert DL. Reduced short interval cortical inhibition correlates with atomoxetine response in children with attention-deficit hyperactivity disorder (ADHD). J Child Neurol. 2014 Dec;29(12):1672-9. doi: 10.1177/0883073813513333. Epub 2014 Jan 10. PMID 24413361
- [Background] Dennis J, White MA, Forrest AD, Yuelling LM, Nogaroli L, Afshari FS, Fox MA, Fuss B. Phosphodiesterase-Ialpha/autotaxin's MORFO domain regulates oligodendroglial process network formation and focal adhesion organization. Mol Cell Neurosci. 2008 Feb;37(2):412-24. doi: 10.1016/j.mcn.2007.10.018. Epub 2007 Nov 12. PMID 18164210
- [Background] Tokumura A, Majima E, Kariya Y, Tominaga K, Kogure K, Yasuda K, Fukuzawa K. Identification of human plasma lysophospholipase D, a lysophosphatidic acid-producing enzyme, as autotaxin, a multifunctional phosphodiesterase. J Biol Chem. 2002 Oct 18;277(42):39436-42. doi: 10.1074/jbc.M205623200. Epub 2002 Aug 9. PMID 12176993
- [Background] Fox MA, Colello RJ, Macklin WB, Fuss B. Phosphodiesterase-Ialpha/autotaxin: a counteradhesive protein expressed by oligodendrocytes during onset of myelination. Mol Cell Neurosci. 2003 Jul;23(3):507-19. doi: 10.1016/s1044-7431(03)00073-3. PMID 12837632
- [Background] Chen YW, Lin HC, Ng MC, Hsiao YH, Wang CC, Gean PW, Chen PS. Activation of mGluR2/3 underlies the effects of N-acetylcystein on amygdala-associated autism-like phenotypes in a valproate-induced rat model of autism. Front Behav Neurosci. 2014 Jun 17;8:219. doi: 10.3389/fnbeh.2014.00219. eCollection 2014. PMID 24987341
- [Background] Mayes DA, Rizvi TA, Titus-Mitchell H, Oberst R, Ciraolo GM, Vorhees CV, Robinson AP, Miller SD, Cancelas JA, Stemmer-Rachamimov AO, Ratner N. Nf1 loss and Ras hyperactivation in oligodendrocytes induce NOS-driven defects in myelin and vasculature. Cell Rep. 2013 Sep 26;4(6):1197-212. doi: 10.1016/j.celrep.2013.08.011. Epub 2013 Sep 12. PMID 24035394
- [Background] Garcia RJ, Francis L, Dawood M, Lai ZW, Faraone SV, Perl A. Attention deficit and hyperactivity disorder scores are elevated and respond to N-acetylcysteine treatment in patients with systemic lupus erythematosus. Arthritis Rheum. 2013 May;65(5):1313-8. doi: 10.1002/art.37893. PMID 23400548
- [Background] Fernandes BS, Dean OM, Dodd S, Malhi GS, Berk M. N-Acetylcysteine in depressive symptoms and functionality: a systematic review and meta-analysis. J Clin Psychiatry. 2016 Apr;77(4):e457-66. doi: 10.4088/JCP.15r09984. PMID 27137430
- [Background] Hardan AY, Fung LK, Libove RA, Obukhanych TV, Nair S, Herzenberg LA, Frazier TW, Tirouvanziam R. A randomized controlled pilot trial of oral N-acetylcysteine in children with autism. Biol Psychiatry. 2012 Jun 1;71(11):956-61. doi: 10.1016/j.biopsych.2012.01.014. Epub 2012 Feb 18. PMID 22342106
- [Background] Berk M, Dean O, Cotton SM, Gama CS, Kapczinski F, Fernandes BS, Kohlmann K, Jeavons S, Hewitt K, Allwang C, Cobb H, Bush AI, Schapkaitz I, Dodd S, Malhi GS. The efficacy of N-acetylcysteine as an adjunctive treatment in bipolar depression: an open label trial. J Affect Disord. 2011 Dec;135(1-3):389-94. doi: 10.1016/j.jad.2011.06.005. Epub 2011 Jun 29. PMID 21719110
- [Background] Fluvoxamine for the treatment of anxiety disorders in children and adolescents. The Research Unit on Pediatric Psychopharmacology Anxiety Study Group. N Engl J Med. 2001 Apr 26;344(17):1279-85. doi: 10.1056/NEJM200104263441703. PMID 11323729
- [Background] Axelrod BN. Validity of the Wechsler abbreviated scale of intelligence and other very short forms of estimating intellectual functioning. Assessment. 2002 Mar;9(1):17-23. doi: 10.1177/1073191102009001003. PMID 11911230
- [Background] Zhu J, Tulsky DS, Price L, Chen HY. WAIS-III reliability data for clinical groups. J Int Neuropsychol Soc. 2001 Nov;7(7):862-6. PMID 11771629
- [Background] Mills KR, Nithi KA. Corticomotor threshold to magnetic stimulation: normal values and repeatability. Muscle Nerve. 1997 May;20(5):570-6. doi: 10.1002/(sici)1097-4598(199705)20:53.0.co;2-6. PMID 9140363
- [Background] Ziemann U. Intracortical inhibition and facilitation in the conventional paired TMS paradigm. Electroencephalogr Clin Neurophysiol Suppl. 1999;51:127-36. No abstract available. PMID 10590943
- [Background] Erkan E, Zhao X, Setchell K, Devarajan P. Distinct urinary lipid profile in children with focal segmental glomerulosclerosis. Pediatr Nephrol. 2016 Apr;31(4):581-8. doi: 10.1007/s00467-015-3239-7. Epub 2015 Nov 4. PMID 26537928
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Result] Doherty AC, Huddleston DA, Horn PS, Ratner N, Simpson BN, Schorry EK, Aschbacher-Smith L, Prada CE, Gilbert DL. Motor Function and Physiology in Youth With Neurofibromatosis Type 1. Pediatr Neurol. 2023 Jun;143:34-43. doi: 10.1016/j.pediatrneurol.2023.02.014. Epub 2023 Mar 3. PMID 36996759

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04481048/Prot_SAP_002.pdf
  • Informed Consent Form (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04481048/ICF_003.pdf